CLINICAL TRIAL: NCT04320927
Title: Iatrogenic Withdrawal Symptoms in Severe Traumatic Brain Injury
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Markus Harboe Olsen, md, Rigshospitalet, Denmark
Other Study IDs: 5798001020855
Record Dates: First submitted 2020-03-23; First posted 2020-03-25 (Actual); Last update posted 2020-04-27 (Actual); Status verified 2020-04

CONDITIONS: Iatrogenic Withdrawal Symptomes

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Iatrogenic withdrawal symptomes has been associated with prolonged mechanical ventilation and the and the derived symptoms such as fever and agitation has been shown to cause significantly prolonged ICU and hospital length of stay. The incidence of IWS in the adult general ICU ranges from 16,7-55%. To this date, the incidence of IWS has not been studied in patients with TBI.

ELIGIBILITY:
Inclusion Criteria:

* adult patients suffering from severe TBI and were mechanical ventilated and received continuous infusions of opioids, benzodiazepines and neuromuscular blocking agents for 72ours or more

Exclusion Criteria:

* age <18 years, patients who died before discharge, chronic alcohol abuse, regular use of heroin, cocaine and amphetamines, chronic use of opioids, patient that were primary admitted to other ICUs and patients that were moved to other ICUs with ongoing infusions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Severe TBI defined as traumatic brain injury that required admission to the neuro-ICU.
Sampling Method: Probability Sample
Enrollment: 215 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-08-01 (Estimated); Study Completion 2020-08-01 (Estimated)

PRIMARY OUTCOMES:
proportion of patients with positive IWS diagnosis | 20-6-2019

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neuroanaesthesiology, Copenhagen, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: No